CLINICAL TRIAL: NCT06170281
Title: A Feasibility Clinical Trial Assessing Patient Preference, Optimum Combinations and Sequences of a Multicomponent, Virtually-Delivered Migraine Behavioral Intervention
Brief Title: Sequential, Multiple Assignment, Double Randomized Preference, Migraine Behavioral Trial
Acronym: SMARTMig
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stanford University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Dr. Yohannes Woldeamanuel, MD, Instructor at Department of Neurology, Stanford University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 70767; K01NS124911 (NIH)
Record Dates: First submitted 2023-10-06; First posted 2023-12-14 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Migraine; Headache; Chronic Migraine; Headache Disorders
Keywords: migraine; headache; behavioral intervention
MeSH Terms: conditions — Migraine Disorders; Headache; Headache Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Random - ME (Active Comparator): participants will be randomized to an intervention involving regular mealtime and regular timed exercise
  Interventions: Behavioral: Migraine Behavioral Treatment
- Random - MS (Active Comparator): participants will be randomized to an intervention involving regular mealtime and regular sleep
  Interventions: Behavioral: Migraine Behavioral Treatment
- Random - SE (Active Comparator): participants will be randomized to an intervention involving regular sleep and regular timed exercise
  Interventions: Behavioral: Migraine Behavioral Treatment
- Choice - ME (Active Comparator): this arm belongs to participants who choose the intervention involving regular mealtime and regular timed exercise
  Interventions: Behavioral: Migraine Behavioral Treatment
- Choice - MS (Active Comparator): this arm belongs to participants who choose the intervention involving regular mealtime and regular sleep
  Interventions: Behavioral: Migraine Behavioral Treatment
- Choice - SE (Active Comparator): this arm belongs to participants who choose the intervention involving regular sleep and regular timed exercise
  Interventions: Behavioral: Migraine Behavioral Treatment

INTERVENTIONS:
Behavioral: Migraine Behavioral Treatment — Migraine Behavioral Treatment involving daily activities

SUMMARY:
This study will unpack the behavioral intervention for migraine and determine the optimum combinations. In addition, the study will test preference and self-selection effects during the trial.

DETAILED DESCRIPTION:
After a 4-week screening period, eligible candidates (14 headache days in 4 week period, with 8 days being migraine) will be randomized into 2 arms -

* Choice Arm: allowed to choose from a menu of migraine behavioral treatment options
* Random: randomized to migraine behavioral treatment options.

After 6 weeks, all participants will be assessed for their migraine frequency. Patients will be considered Responders if the migraine frequency is reduced to 50%. The Non-responders (NR) of the Choice Arm will be again given a chance to pick any of the 3 arms. The NR of the randomized arm will be randomized to any of the 3 arms. The responders will continue for 6 more weeks in their original arms. By the end of the 12 weeks, all participants will complete the study, and migraine frequency will be compared between the different groups. All behavioral interventions will be delivered virtually.

ELIGIBILITY:
Inclusion Criteria:

* have chronic migraine for a minimum of 1-year
* aged 18 years and older

Exclusion Criteria:

* secondary headache disorders
* children younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility in terms of recruitment and adherence rates | 12 weeks
  recruitment rate, adherence rate

SECONDARY OUTCOMES:
Migraine Frequency | at baseline 4 weeks before randomization, week 2-6 after date of randomization, week 8-12 after date of randomization
  migraine day frequency
Headache Self-efficacy | at baseline 4 weeks before randomization, week 2-6 after date of randomization, week 8-12 after date of randomization
  headache self-efficacy measured using validated headache self-efficacy questionnaire
Migraine Intensity | at baseline 4 weeks before randomization, week 2-6 after date of randomization, week 8-12 after date of randomization
  migraine intensity, self-reported

CONTACTS AND LOCATIONS:
Overall Officials: Yohannes W Woldeamanuel, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: starting 6 months after publication, for 2 years
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).

REFERENCES:
- [Background] Woldeamanuel YW, Sanjanwala BM, Peretz AM, Cowan RP. Exploring Natural Clusters of Chronic Migraine Phenotypes: A Cross-Sectional Clinical Study. Sci Rep. 2020 Feb 18;10(1):2804. doi: 10.1038/s41598-020-59738-1. PMID 32071349
- [Background] Woldeamanuel YW, Cowan RP. The impact of regular lifestyle behavior in migraine: a prevalence case-referent study. J Neurol. 2016 Apr;263(4):669-76. doi: 10.1007/s00415-016-8031-5. Epub 2016 Jan 25. PMID 26810728
- [Background] Woldeamanuel YW, Blayney DW, Jo B, Fisher SE, Benedict C, Oakley-Girvan I, Kesler SR, Palesh O. Headache outcomes of a sleep behavioral intervention in breast cancer survivors: Secondary analysis of a randomized clinical trial. Cancer. 2021 Dec 1;127(23):4492-4503. doi: 10.1002/cncr.33844. Epub 2021 Aug 6. PMID 34357593